CLINICAL TRIAL: NCT00882726
Title: A Phase 1, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Ascending Intravenous and Subcutaneous Single-Dose Study in Healthy Subjects and Ascending Subcutaneous Multiple-Dose Study in Subjects With Type 2 Diabetes Mellitus to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immune Response of CNTO 3649
Brief Title: A Study of the Safety, Pharmacokinetics, and Pharmacodynamics of CNTO 3649 in Healthy Adults and Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015562; CNTO3649DIB1001 (Other: Centocor)
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; CNTO 3649; safety; Phase I; healthy adults; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CNTO 3649 IV (Healthy participants) (Experimental)
  Interventions: Drug: CNTO 3649 IV (Healthy participants); Drug: Placebo
- CNTO 3649 SC (Healthy participants) (Experimental)
  Interventions: Drug: CNTO 3649 SC (Healthy participants); Drug: Placebo
- CNTO 3649 SC (Diabetic patients) (Experimental)
  Interventions: Drug: CNTO 3649 SC (Diabetic patients); Drug: Placebo

INTERVENTIONS:
Drug: CNTO 3649 IV (Healthy participants) — Healthy participants will each receive a single dose of CNTO 3649 (1, 3, 10, 30, 100 or 300 microgram per kilogram, subject to change) as a 2-hour IV infusion.
  Arms: CNTO 3649 IV (Healthy participants)
Drug: CNTO 3649 SC (Healthy participants) — Healthy participants will each receive a single dose of CNTO 3649 (10, 30, 100 or 300 microgram per kilogram, subject to change) as a SC injection.
  Arms: CNTO 3649 SC (Healthy participants)
Drug: CNTO 3649 SC (Diabetic patients) — Diabetic patients will receive multiple doses of CNTO 3649 (30, 100 or 300 microgram per kilogram, subject to change) as subcutaneous injections once weekly for 4 consecutive weeks.
  Arms: CNTO 3649 SC (Diabetic patients)
Drug: Placebo — Participants within each dosing group who are randomized to placebo will receive a corresponding IV infusion or SC injection of placebo.

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and pharmacodynamics of CNTO 3649 following a single dose in healthy adults and following multiple doses in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), placebo controlled, double-blind (neither physician nor patient knows the name of the assigned study medication), ascending-dose study to assess the safety, tolerability, immune response, pharmacokinetics (what the body does to the drug), and pharmacodynamics (what the drug does to the body) of CNTO 3649. The study population will consist of approximately 80 healthy participants (Part 1) and approximately 36 type 2 diabetic patients (Part 2). All participants will be randomized to CNTO 3649 or placebo in the ratio of 3:1. Out of 80 healthy participants, 48 participants will receive single doses of CNTO 3649 (6 dose levels) or placebo as an intravenous infusion (directly into a vein) and 32 participants will receive single doses of CNTO 3649 (4 dose levels) or placebo as a subcutaneous (under the skin) injection. All 36 diabetic patients will receive multiple doses of CNTO 3649 (3 dose levels) or placebo as subcutaneous injections. There will be a screening period of 30 days and 45 days for healthy participants and diabetes patients, respectively. Healthy participants will be in the study for 9 weeks. Diabetic patients will be in the study for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 (healthy participants): Demonstrate an understanding of the study and sign an informed consent form
* Healthy male or female subjects with no clinically relevant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments including complete blood count, coagulation tests, urinalysis, measurement of vital signs, and ECG
* Age 18 to 55
* Have a body mass index (BMI) of 18.5 to 30 kg/m2 and weight of 50 to 100 kg
* Part 2 (patients with type 2 diabetes): Type 2 Diabetic male or female subjects diagnosed at least 12 months prior to screening and are stably managed for >= 3 months
* HbA1c levels within the range of 6% to 10% if being treated with diet and exercise alone, and 6% to 9% if on therapy
* BMI 18.5 to 37 kg/m2. Age 18 to 65 years.

Exclusion Criteria:

* Part 1 (healthy participants): Currently have or have a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the subject
* Part 2 (patients with type 2 diabetes): Any clinically significant medical illness or medical disorders (with the exception of diagnosis of T2DM, well-controlled hypertension, or well-controlled dyslipidemia) the investigator considers should exclude the subject. History of more than 3 days of insulin use in the last 3 months, or any thiazolidinedione medications, any alpha glucosidase inhibitors, or exenatide within 3 months of the screening visit. History of clinically significant acute or chronic diabetic complications. History of severe hypoglycemic reaction in the 6 months prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single IV or SC administration of CNTO 3649 in healthy participants; Safety and tolerability of multiple SC injections of CNTO 3649 in Type 2 Diabetic Patients | Week 1 to Week 5 (for healthy participants) and Week 1 to Week 8 (for diabetic patients)

SECONDARY OUTCOMES:
Pharmacokinetics, pharmacodynamics and immunogenicity of CNTO 3649 following single and multiple administrations. | Week 1 to Week 5 (for healthy participants) and Week 1 to Week 8 (for diabetic patients)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Clinical Trial, Study Director — Centocor, Inc.
Locations (3):
- United States (3):
  - Miramar, Florida
  - San Antonio, Texas
  - Tacoma, Washington

REFERENCES:
- See also: A Study of the Safety, Pharmacokinetics, and Pharmacodynamics of CNTO 3649 in Healthy Adults and Patients With Type 2 Diabetes Mellitus. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=189&filename=CR015562_CSR.pdf